CLINICAL TRIAL: NCT06259058
Title: Evaluate the Efficacy and Safety of Stereotactic Body Radiation Therapy Followed by NALIRIFOX vs NALIRIFOX for Borderline Resectable Pancreatic Cancer: a Phase Ib/II, Multicenter, Open-label Trial
Brief Title: Stereotactic Body Radiation Therapy Followed by NALIRIFOX vs NALIRIFOX for Borderline Resectable Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-PC-K04
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer
Keywords: borderline resectable; NALIRIFOX; stereotactic body radiation therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NALIRIFOX + SBRT + NALIRIFOX + Surgery + NALIRIFOX (Experimental): Patients receive 3 cycles of NALIRIFOX followed by SBRT (30Gy/5Fx). Then undergo surgery and receive 6 cycles of NALIRIFOX after surgery. NALIRIFOX consists of irinotecan liposome injection, oxaliplatin, 5 FU/LV.
  Interventions: Drug: Irinotecan liposome injection; Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Leucovorin; Radiation: SBRT
- NALIRIFOX + Surgery + NALIRIFOX (Active Comparator): Patients receive 6 cycles of NALIRIFOX. Then undergo surgery and receive 6 cycles of NALIRIFOX after surgery. NALIRIFOX consists of irinotecan liposome injection, oxaliplatin, 5 FU/LV.
  Interventions: Drug: Irinotecan liposome injection; Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Irinotecan liposome injection — 50 mg/m² on Day 1 of a 14-day cycle
  Other Names: Nal-IRI
Drug: Oxaliplatin — 60 mg/m² on Day 1 of a 14-day cycle
  Other Names: Eloxatin
Drug: 5-Fluorouracil — 2400 mg/m² continuous IV infusion in 46 h
  Other Names: 5-FU; flurouracil; Adrucil
Drug: Leucovorin — 400 mg/m² on Day 1 of a 14-day cycle
  Other Names: Folinic Acid
Radiation: SBRT — 30Gy/5Fx
  Arms: NALIRIFOX + SBRT + NALIRIFOX + Surgery + NALIRIFOX

SUMMARY:
This multicentric open-label trial will compare the efficacy and safety of stereotactic body radiation therapy (SBRT) followed by NALIRIFOX (5-fluorouracil, leucovorin, irinotecan liposome injection and oxaliplatin) vs NALIRIFOX for borderline resectable pancreatic cancer (BRPC).

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy or chemoradiotherapy can increase the R0 resection rate and improve survival in BRPC. However, there is no standard treatment regimen. The National Comprehensive Cancer Network (NCCN) guidelines recommend FOLFIRINOX (irinotecan + oxaliplatin +5-FU/LV) and FOLFIRINOX+ chemoradiotherapy for PDAC neoadjuvant treatment.

Liposomal irinotecan is a new pharmaceutical form of traditional irinotecan. It adopts a special loading technology to encapsulate traditional irinotecan in liposomes, which can avoid its hydrolysis under physiological conditions, increase the affinity with cancer cells, overcome drug resistance, increase the drug uptake by cancer cells, reduce the drug dose,improve the efficacy and reduce the toxic side effects. The aim of this study is to compare the efficacy and safety of NALIRIFOX + surgery + NALIRIFOX or surgery + NALIRIFOX in high-risk patients with resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old.
* Histologically or cytologically proven pancreatic ductal adenocarcinoma.
* Multidisciplinary assessment as borderline resectable disease.
* At least one measurable lesion (according to RECIST v1.1).
* No prior antitumor therapy for pancreatic cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 1.
* The expected survival time ≥3 months.
* Adequate bone marrow function as evidenced by: 1) Absolute neutrophil count (ANC) ≥1.5×10^9/L, 2) Platelet count ≥100×10^9/L, 3) Hemoglobin (Hb) ≥90 g/L, 4) White blood cell (WBC) ≥3.0×10^9/L.
* Adequate hepatic function as evidenced by: 1) Serum total bilirubin ≤1.5 × upper limit of normal (ULN), 2) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN
* Adequate renal function as evidenced by serum creatinine (Cr)≤1.5 × ULN or creatinine clearance ≥60 mL/min.
* Agree and be able to comply with the plan during the study period. Provide written informed consent before entering the study screening.

Exclusion Criteria:

* Any other malignancy within 5 years, with the exception of cured in-situ carcinoma or basal cell carcinoma etc.
* Patients with distant metastases and/or cannot complete resection.
* Active, uncontrolled bacterial, viral, or fungal infections that require systemic treatment.
* Active HIV, HBV, HCV infection.
* Combined with uncontrollable systemic diseases.
* Presence of severe gastrointestinal disease (including active bleeding, > grade 1 obstruction [CTCAE v5.0], or > grade 1 diarrhea [CTCAE v5.0]).
* History of allergy or hypersensitivity to drug or any of their excipients.
* Patients who have chemotherapy and surgery contraindications.
* Documented serum albumin ≤3 g/dL
* Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1 within 14 days before the first administration.
* Pregnant or breastfeeding women, or subjects of childbearing age who refuse contraception.
* Participated in other trial within 30 days before the first administration.
* Patients who are not suitable to participate in this trial for any reason judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 4 months
  Defined as the proportion of patients who have achieved R0 resection.

SECONDARY OUTCOMES:
Objective Response Rate | 3 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1
Surgical Conversion Rate (R0 / R1 resection) | 4 months
  Defined as the percentage of patients that underwent a R0/R1 resection.
Tumor regression grade | 4 months
  The classification is mainly based on the proportion of residual tumors and fibrosis in the primary tumor, used to evaluate the patient's response to neoadjuvant therapy and predict prognosis.
Event-free Survival | 1 year
  Defined as the time between signing the informed consent form to the first documentation of 1) disease progression (local recurrence, new lesions or distant metastasis), 2) a second malignant tumor occurs, or 3) death due to any cause.
Overall survival | 2 years
  Defined as the time between signing the informed consent form and death due to various causes.
Incidence of adverse events | 7 months
  Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Professor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital

IPD SHARING:
Plan to Share IPD: No